CLINICAL TRIAL: NCT01339741
Title: The Efficacy of Vitamin D3 for the Treatment of Chronic Plaque Type Psoriatic Patients With Vitamin D Deficiency and Insufficiency: a Randomized Controlled Trial
Brief Title: Efficacy of Vitamin D3 for the Treatment of Psoriatic Patients With Vitamin D Deficiency and Insufficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Chotinij Lertphanichkul, M.D., Faculty of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PsoriasisVitaminD; COA No. 057/2011 (Other: Faculty of Medicine, Chulalongkorn University)
Record Dates: First submitted 2011-04-20; First posted 2011-04-21 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Psoriasis Vulgaris; Vitamin D Deficiency
Keywords: Psoriasis Vulgaris; Vitamin D Deficiency; Vitamin D Insufficiency; Vitamin D Supplement; Psoriasis Area and Severity Index (PASI Score); Dermatologic Life Qualify Index (DLQI)
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Vitamin D (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3, oral supplement, 12 weeks
  Arms: Vitamin D
Drug: Placebo — Placebo, oral route, 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this research is to study whether vitamin D supplement can improve clinical outcome (PASI score) in psoriasis vulgaris with vitamin D insufficiency and deficiency.

DETAILED DESCRIPTION:
While psoriasis is not a lethal disease, the disease itself can impact patients' quality of life. Nowadays there are several researches on vitamin D functions. Recently review article of vitamin D deficiency by Holick MF., stated that vitamin D can play a role in decreasing the risk of osteoporosis and other chronic diseases such as malignancy, autoimmune disease, infectious disease, cardiovascular disease, and psoriasis. Moreover, vitamin D effects on keratinocyte by decreasing abnormal cell proliferation, differentiation, apoptosis and controlling immunological process via the suppression of T-cell activation, regulation of cytokine secretion patterns, induction of regulatory T-cell, modulation of T-cell proliferation and interference with T-cell apoptosis.

Thus, our objective is to look for other alternative treatment, which may have less side effects and acceptable clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderately severe (PASI ≤ 10), chronic plaque type psoriasis vulgaris patient, who is a new case or has at least treatment-free period as following: 4 weeks for topical calcipotriol, topical corticosteroid or 8 weeks for systemic therapy (i.e. cyclosporine, acitretin, methotrexate) or 12 weeks for Psoralen Ultraviolet A (PUVA), phototherapy or biological treatment.
* Age 18-year-old to 70-year-old.
* Psoriasis vulgaris patient with vitamin D insufficiency or deficiency.

Exclusion Criteria:

* Pregnancy or Lactating mother.
* Subject with history of major gastrointestinal surgery or gastric bypass surgery.
* Subject with history of pustular psoriasis.
* Subject with active psoriatic arthritis.
* Subject with prior phototherapy within the past 3 months.
* Subject with history of hypocholesterolemia (serum cholesterol < 120 mg/dl) or primary hyperparathyroidism.
* Subject who regularly takes vitamin D supplement exceed 3,000 iu/day and high vitamin D diet, for example cod liver oil.
* Subject with liver disease, cystic fibrosis, Crohn's disease, celiac sprue, renal disease, pancreatic disease, and inflammatory bowel disease.
* Subject taking following medication: corticosteroid, orlistat, rifampicin, isoniazid, ketoconazole, statin, and cholestyramine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI Score) | 12 weeks
  Normal vitamin D level after replacement correlate with improved clinical outcome (PASI Score) of psoriasis vulgaris.

SECONDARY OUTCOMES:
Dermatologic Life Qualify Index (DLQI) | 12 weeks
  Normal vitamin D level after replacement correlates with better DLQI.

CONTACTS AND LOCATIONS:
Overall Officials: Chotinij Lertphanichkul, M.D., Principal Investigator — Chulalongkorn University
Locations (1):
- Chotinij Lertphanichkul, M.D., Patumwan, Bangkok, Thailand

REFERENCES:
- [Background] Griffiths CE, Barker JN. Pathogenesis and clinical features of psoriasis. Lancet. 2007 Jul 21;370(9583):263-271. doi: 10.1016/S0140-6736(07)61128-3. PMID 17658397
- [Background] Kurd SK, Troxel AB, Crits-Christoph P, Gelfand JM. The risk of depression, anxiety, and suicidality in patients with psoriasis: a population-based cohort study. Arch Dermatol. 2010 Aug;146(8):891-5. doi: 10.1001/archdermatol.2010.186. PMID 20713823
- [Background] Choi J, Koo JY. Quality of life issues in psoriasis. J Am Acad Dermatol. 2003 Aug;49(2 Suppl):S57-61. doi: 10.1016/s0190-9622(03)01136-8. PMID 12894127
- [Background] Menter A, Gottlieb A, Feldman SR, Van Voorhees AS, Leonardi CL, Gordon KB, Lebwohl M, Koo JY, Elmets CA, Korman NJ, Beutner KR, Bhushan R. Guidelines of care for the management of psoriasis and psoriatic arthritis: Section 1. Overview of psoriasis and guidelines of care for the treatment of psoriasis with biologics. J Am Acad Dermatol. 2008 May;58(5):826-50. doi: 10.1016/j.jaad.2008.02.039. PMID 18423260
- [Background] Hosomi J, Hosoi J, Abe E, Suda T, Kuroki T. Regulation of terminal differentiation of cultured mouse epidermal cells by 1 alpha,25-dihydroxyvitamin D3. Endocrinology. 1983 Dec;113(6):1950-7. doi: 10.1210/endo-113-6-1950. PMID 6196178
- [Background] Morimoto S, Kumahara Y. A patient with psoriasis cured by 1 alpha-hydroxyvitamin D3. Med J Osaka Univ. 1985 Mar;35(3-4):51-4. No abstract available. PMID 4069059
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Soontrapa S, Soontrapa S, Bunyaratavej N, Rojanasthien S, Kittimanon N, Lektrakul S. Vitamin D status of Thai premenopausal women. J Med Assoc Thai. 2009 Sep;92 Suppl5:S17-20. PMID 19891376
- [Background] Su MJ, Bikle DD, Mancianti ML, Pillai S. 1,25-Dihydroxyvitamin D3 potentiates the keratinocyte response to calcium. J Biol Chem. 1994 May 20;269(20):14723-9. PMID 7910167
- [Background] Bikle DD, Pillai S. Vitamin D, calcium, and epidermal differentiation. Endocr Rev. 1993 Feb;14(1):3-19. doi: 10.1210/edrv-14-1-3. No abstract available. PMID 8491153
- [Background] Rigby WF, Stacy T, Fanger MW. Inhibition of T lymphocyte mitogenesis by 1,25-dihydroxyvitamin D3 (calcitriol). J Clin Invest. 1984 Oct;74(4):1451-5. doi: 10.1172/JCI111557. PMID 6332829
- [Background] Boonstra A, Barrat FJ, Crain C, Heath VL, Savelkoul HF, O'Garra A. 1alpha,25-Dihydroxyvitamin d3 has a direct effect on naive CD4(+) T cells to enhance the development of Th2 cells. J Immunol. 2001 Nov 1;167(9):4974-80. doi: 10.4049/jimmunol.167.9.4974. PMID 11673504
- [Background] Penna G, Adorini L. 1 Alpha,25-dihydroxyvitamin D3 inhibits differentiation, maturation, activation, and survival of dendritic cells leading to impaired alloreactive T cell activation. J Immunol. 2000 Mar 1;164(5):2405-11. doi: 10.4049/jimmunol.164.5.2405. PMID 10679076
- [Background] May E, Asadullah K, Zugel U. Immunoregulation through 1,25-dihydroxyvitamin D3 and its analogs. Curr Drug Targets Inflamm Allergy. 2004 Dec;3(4):377-93. doi: 10.2174/1568010042634596. PMID 15584887
- [Background] Reichrath J. Vitamin D and the skin: an ancient friend, revisited. Exp Dermatol. 2007 Jul;16(7):618-25. doi: 10.1111/j.1600-0625.2007.00570.x. PMID 17576242
- [Background] Bikle D. Nonclassic actions of vitamin D. J Clin Endocrinol Metab. 2009 Jan;94(1):26-34. doi: 10.1210/jc.2008-1454. Epub 2008 Oct 14. PMID 18854395
- [Background] Kragballe K, Wildfang IL. Calcipotriol (MC 903), a novel vitamin D3 analogue stimulates terminal differentiation and inhibits proliferation of cultured human keratinocytes. Arch Dermatol Res. 1990;282(3):164-7. doi: 10.1007/BF00372616. PMID 2164359
- [Background] Bagot M, Charue D, Lescs MC, Pamphile RP, Revuz J. Immunosuppressive effects of 1,25-dihydroxyvitamin D3 and its analogue calcipotriol on epidermal cells. Br J Dermatol. 1994 Apr;130(4):424-31. doi: 10.1111/j.1365-2133.1994.tb03373.x. PMID 8186106
- [Background] Bruce S, Epinette WW, Funicella T, Ison A, Jones EL, Loss R Jr, McPhee ME, Whitmore C. Comparative study of calcipotriene (MC 903) ointment and fluocinonide ointment in the treatment of psoriasis. J Am Acad Dermatol. 1994 Nov;31(5 Pt 1):755-9. doi: 10.1016/s0190-9622(94)70237-3. PMID 7929921
- [Background] Morimoto S, Yoshikawa K, Kozuka T, Kitano Y, Imanaka S, Fukuo K, Koh E, Kumahara Y. An open study of vitamin D3 treatment in psoriasis vulgaris. Br J Dermatol. 1986 Oct;115(4):421-9. doi: 10.1111/j.1365-2133.1986.tb06236.x. PMID 3022784